CLINICAL TRIAL: NCT06504784
Title: Effect of Dietary Fiber on Gut Microbiota Composition and Immune Response to Influenza Vaccination in Ulcerative Colitis Patients on Immunosuppressive Therapy: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Role of Gut Bacteria in the Immune Response to Vaccination in Patients With Ulcerative Colitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Calmino group AB (Unknown)
Responsible Party: Principal Investigator, Jóhann P. Hreinsson, MD, PhD, associate professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PreVac2023
Record Dates: First submitted 2024-06-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: Randomization and Concealed allocation will be assured by the distribution of investigational products by a nurse/researcher at the unit, otherwise not involved in the conduct of the study. The randomization schedule will be kept in a locked cabinet until the completion of the trial and all data had been entered into a computer database. Both the investigators and the participants will be blinded to treatment arm assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Fibre Mixture (Experimental): Study participants receive 10g/day of dietary fibre mixture (a mixture of oligo-and polysaccharides), divided into two doses and administered orally for 6 weeks.
  Interventions: Dietary Supplement: Dietary Fiber Mixture
- Placebo (Placebo Comparator): Study participants receive 10g/day of placebo (glucose) matching the fibre mixture in colour and flavor, divided into two doses and administered orally for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Fiber Mixture — 10g/day of dietary fibre mixture - a mixture of oligo-and polysaccharides
  Arms: Dietary Fibre Mixture
Other: Placebo — 10g/day of placebo (glucose)
  Arms: Placebo

SUMMARY:
Patients with the inflammatory bowel disease ulcerative colitis (UC) are a high-risk group encouraged to get vaccinated against seasonal influenza. It is also known that UC patients may have an altered gut microbiota.

Patients with more severe disease are treated with immunosuppressive medications such as thiopurines and biologics that block pro-inflammatory cytokines. However, these treatments makes patients more susceptible to infections and results in a poorer response to certain types of vaccinations, as the immunosuppressive treatment aims to suppress mechanisms in the immune response.

The purpose of the study is to determine if dietary fibers can improve the immune response to influenza vaccination in UC patients treated with immunosuppressive medications. Further, the study aims to determine if dietary fibers (prebiotics) can enrich the composition and function of the gut microbiota in UC patients.

DETAILED DESCRIPTION:
Project Description:

The purpose of the study is to determine if dietary fibers can improve the immune response to influenza vaccination in UC patients treated with immunosuppressive medications. The investigators also intend to determine if dietary fibers (prebiotics) can enrich the composition and function of the gut microbiota in UC patients.

Background and Justification:

Patients with moderate to severe UC often require lifelong medical treatment. Long-term treatment typically includes medications such as 5-ASA, immunomodulatory agents like thiopurines, and/or antibodies or biologics that block pro-inflammatory cytokines. These medical treatments aim to suppress the patient's inflammatory activity both systemically and locally in the gut. The treatment is often effective, leading to complete or partial healing of gut inflammation, known as remission. Unfortunately, the treatment also makes patients more susceptible to infections and results in a poorer response to certain types of vaccinations.

Patients with UC are a high-risk group and are encouraged to vaccinate against the seasonal influenza virus. Vaccination activates immune cells to produce antibodies that protect against the influenza virus. The effectiveness of the vaccination is measured by the levels (titers) of influenza-specific antibodies formed. Previous studies have shown that patients treated with biologics such as antibodies against the pro-inflammatory cytokine TNF, have a poorer response to various vaccinations, including influenza, and therefore receive less protection against the infection.

Recent studies have shown that the composition of the gut microbiota at the time of vaccination affects the response/protection from vaccination in healthy volunteers. The studies also implicate research subjects with a "poorer"/more depleted composition of gut bacteria with a reduced ability to form antibodies and thus create immunological protection in response to vaccination. It is known that UC patients have a depleted composition of gut bacteria compared to healthy individuals.

Previous studies have suggested that it may be possible to improve the composition of gut bacteria in UC patients by enriching the diet with dietary fibers, known as prebiotics, which promote the presence of certain gut bacteria believed to have health-promoting effects. There are many different types of dietary fibers consisting of carbohydrates and starch. Examples of dietary fibers include inulin, mannose, galacto-oligosaccharides, and starch.

Study Design:

Recruitment of Participants:

UC Patients: Patients treated at the Gastroenterology Clinic, Sahlgrenska University Hospital, will be invited via mail and follow-up phone calls. This study aims to recruit 100 patients (18-65 years) on maintenance treatment with anti-TNF agents and/or thiopurines, or 5-ASA.

Healthy subjects: Recruited through local advertising at Sahlgrenska University Hospital and social media. This study aims to recruit 50 healthy participants as control (18-65 years).

All research subject will be informed and asked verbally to participate in the study. Those who agree will sign informed consent.

Intervention:

All study participants will be randomized to receive either 10 g of dietary fiber per day (divided into 2 doses) or 10 g of placebo (glucose, divided into 2 doses) for 3 weeks before the influenza vaccination. They will continue to take dietary fiber or placebo for 3-4 weeks after the vaccination.

The dietary fiber mix (total 10 g/day) includes inulin, acetylated polymannose, galacto-oligosaccharides, and resistant starch. Intervention products were provided by Calmino group AB, Sweden.

All research subjects will be vaccinated after 3 weeks of intervention period. The vaccination procedure and dosage will be the same as in standard clinical practice.

All participants will complete questionnaires to assess GI symptom severity, and blood and fecal samples will be collected at baseline, 3 weeks after intervention (vaccination visit), 6 weeks after intervention/end of intervention (3 weeks post-vaccination) and at long term follow-up ( 20-25 weeks post-vaccination).

Significance:

This is the first time the impact of dietary fibers on vaccination response is being studied in UC patients treated with anti-inflammatory drugs. If the study shows favorable results, it could lead to changes in clinical practice, including advising patients to intake dietary fiber to enrich gut flora, improve immune response, and enhance protection during vaccination.

ELIGIBILITY:
Inclusion Criteria:

* UC patients, aged 18-65, in remission, with stable maintenance treatment for at least 6 months consisting of anti-TNF medications and/or thiopurines, or 5-ASA.
* Healthy volunteers, aged 18-65.

Exclusion Criteria:

* Comorbidity according to the Charlston Comorbidity Index
* Ongoing immunosuppressive treatment for a condition other than inflammatory bowel disease
* Colorectal surgical treatment for inflammatory bowel disease
* Treatment with antibiotics in the past 3 months
* Intake of probiotic or prebiotic dietary supplements in the past 3 months
* Inability to understand information about the study or provide informed consent

Additional Exclusion Criteria for Healthy Volunteers:

-Inflammatory bowel disease or suspicion thereof

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The level of influenza-specific antibodies (titers) in blood samples measured post-vaccination. | Measured at Visit 2 (day of vaccination), Visit 3 (3-4 weeks post-vaccination), and Visit 4 (20-25 weeks post-vaccination).
  The level of influenza-specific antibodies (titers) in blood samples of UC patients measured post-vaccination in intervention group (receiving dietary fiber) compared to patients in the placebo group.
Effect of Dietary Fibers on Gastrointestinal Symptoms using the validated Gastrointestinal Symptom Rating Scale (GSRS) questionnaire in Patients with Ulcerative Colitis comparing baseline vs. end of 6 week oral intervention with dietary fiber. | GI symptoms using GSRS symptom questionnaire were assessed at baseline and at 3 week and 6 weeks after intervention
  GI symptoms are assessed using the validated Gastrointestinal Symptom Rating Scale (GSRS). GSRS is a 15 item measure of IBS symptom severity. The scale measures the severity of each symptom on a scale from 1 to 7. Maximum total score is 7 and minimum score is 1, where a higher score indicates higher gastrointestinal symptom severity.
Effect of Dietary Fibers on disease activity assessed using a modified Mayo score form in Patients with Ulcerative Colitis comparing baseline vs. end of 6 week oral intervention. | Mayo score (modified) will be measured at baseline and at 3 week and 6 weeks after intervention
  Disease activity is assessed using a modified Mayo score (UC patients only). Mayo score measures disease activity on a scale from to 6, where the maximum score is 6 and minimum score is 0, and higher score indicated worse outcome with regards to disease activity. Change in total Mayo score will be evaluated.

SECONDARY OUTCOMES:
Effect of dietary fiber intake on metabolite composition in UC patients and healthy controls comparing baseline vs. end of 6 week oral intervention. | Analyzed from fecal samples collected at Visit 1 (baseline), Visit 2 (day of vaccination), Visit 3 (3-4 weeks post-vaccination), and Visit 4 (20-25 weeks post-vaccination).]
  Change in metabolite profile/composition in UC patients and healthy controls after intervention with dietary fiber compared to placebo will be established. Fecal samples will be used to evaluate the Metabolite profile using untargeted Liquid chromatography coupled to a mass spectrometer (LC-MS). Change in the metabolite profile measured as metabolite signal response from Baseline to 6 Weeks after intervention will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No